CLINICAL TRIAL: NCT04924764
Title: Prediction of Recovery in Patients With Neck Pain: Prospective Longitudinal Study
Brief Title: Prediction of Recovery in Patients With Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/0876 Seerat Rashid
Record Dates: First submitted 2021-05-19; First posted 2021-06-14 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Neck Pain; Chronic Neck Pain; Cervical Radiculopathy
Keywords: Prediction Model; neck pain; recovery; chronic; sub acute
MeSH Terms: conditions — Neck Pain; Radiculopathy; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follow-up on daily basis (Active Comparator): Patient receiving treatments on daily basis (5 days a week)
  Interventions: Other: Conventional physical therapy.
- Follow-up on alternate days (Active Comparator): Patients receiving treatment on alternate days (3 days a week)
  Interventions: Other: Conventional physical therapy.

INTERVENTIONS:
Other: Conventional physical therapy. — Conventionally used intervention for subacute and chronic neck pain.

SUMMARY:
This prognostic prediction model will be a reference for the health care professionals in clinical decision making and subsequent outcomes in dealing with patients having sub-acute and chronic neck pain, as well as, it will be a guide regarding therapeutic management and patients' education. Although various studies have evaluated the prognostic factors for individual neck pain conditions or treatment, to author Knowledge, no such prognostic model is available yet that predict the recovery in patients of sub-acute and chronic neck pain when managed conservatively. Therefore, this study is aimed to create a prediction model suggesting the recovery time for neck pain.

DETAILED DESCRIPTION:
Neck pain is a highly prevalent condition that leads to considerable pain, disability, and economic cost. It not only constitutes a major personal burden but also affects families, the health system and the economic structure of countries. Neck pain is described as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage" in the neck region, which starts at the superior nuchal line and continues down to the level of the scapular spine. Acute, sub-acute and chronic neck pain is defined as neck pain with full-time sick-listing for 0 - 21 days (3 weeks), 22 - 84 days (4-12 weeks) and more than 12 weeks, respectively. A number of studies have explored prognostic factors for neck pain. Most frequently reported prognostic factors are age, gender, pain severity, a history of neck pain, concomitant low back pain, duration of pain, occupation, previous trauma, and degenerative changes on X-ray. Physiotherapy interventions for chronic neck pain showing the strongest support for an effect on pain are strength and endurance training. Two of the most widely used treatment strategies for the management of neck pain is exercise therapy (ET) and manual therapy (MT). ET is defined as a regimen or plan of physical activities designed and prescribed for any therapeutic goals, which includes strength exercises, stabilization exercises and endurance exercises. MT may is defined as "the use of hands to apply a force with therapeutic intent. various studies have evaluated the prognostic factors for individual neck pain conditions or treatment. but the author Knowledge, no such prognostic model is available yet that predict the recovery in patients of sub-acute and chronic neck pain when managed conservatively.

ELIGIBILITY:
Inclusion Criteria:

* Subacute and chronic neck pain.
* Patients with neck pain with a score of 4-10 on the numeric pain rating scale.

Exclusion Criteria:

* Acute neck pain.
* Neck pain due to fracture, tumour, infection or metabolic bone disease.
* History of cervical spine injury or surgery.
* Patients presented with disc herniation.
* Cervical instability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | Up to 2 months
  The Numeric pain rating scale (NPRS) is a self-reported, or clinician-administered, measurement tool consisting of a numerical point scale with extreme anchors of 'no pain' to 'extreme pain. The scale is typically set up on a horizontal or vertical line, ranges most commonly from 0-10 or 0-100, and can be administered in written or verbal form. The patient is asked to rate his/her pain intensity and a particular time frame or descriptor is established (e.g. within the last 24 h, today, worst pain, average pain, or least pain). The NPRS scores are high on ease of administration and simplicity for scoring. The last reading will be taken when the NPRS score will be less than 3.
Neck disability index | Up to 2 months
  The Neck Disability Index (NDI) is a 10-item questionnaire that measures a patient's self-reported neck pain-related disability. The NDI is the most widely used, translated and oldest questionnaire for neck pain. Questions include activities of daily living, such as personal care, lifting, reading, work, driving, sleeping, recreational activities, pain intensity, concentration and headache. Each question is measured on a scale from 0 (no disability) to 5, and an overall score out of 100 is calculated by adding each item score together and multiplying it by two. A higher NDI score means the greater a patient's perceived disability due to neck pain. The "minimally clinically important change" by patients has been found to be 5 or 10%. The last reading will be taken when the NPRS score will be less than 3.
Range of Motion | Up to 2 months
  Goniometric measurements are used by physical therapists to quantify baseline limitations of motion, decide on appropriate therapeutic interventions, and document the effectiveness of these interventions. Goniometry can be considered a fundamental part of the "basic science" of physical therapy. To most physical therapists, however, the universal goniometer (i.e. full-circle manual goniometer) remains the most versatile and widely used instrument in clinical practice. The last reading will be taken when the NPRS score will be less than 3.
Manual muscle testing for strength of cervical muscle | Up to 2 months
  Medical Research Council Manual Muscle Testing scale is the most commonly accepted method of evaluating muscle strength. This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly; 0 means no muscle activation, 1 means trace muscle activation, such as a twitch, without achieving full Range of Motion (ROM), 2 means muscle activation with gravity eliminated, achieving full ROM, 3 means muscle activation against gravity, full ROM, 4 means muscle activation against some resistance, full ROM, 5 means muscle activation against examiner's full resistance, full ROM. The last reading will be taken when the NPRS score will be less than 3.

SECONDARY OUTCOMES:
Pain Anxiety symptom scale | Up to 2 months
  The Pain Anxiety symptom scale -20 (PASS-20) was constructed by extracting 20 items from its 40-item parent measure Pain Anxiety symptom scale (PASS) (18). The PASS-20 is a 20-item self-report instrument, measuring 4 factorially distinct components of pain-related anxiety. The cognitive subscale assesses cognitive anxiety symptoms, such as racing thoughts and impaired concentration due to pain. The fear subscale assesses fearful thoughts and anticipated negative consequences of pain. The escape/avoidance subscale assesses behavioural responses that reduce or terminate pain. The physiological anxiety subscale assesses physiological arousal in response to pain. Each item is rated on a 6-point Likert scale ranging from 0 (never) to 5 (always). Summing each subscale provides a score that can be considered a general measure of pain-related anxiety. The last reading will be taken when the NPRS score will be less than 3.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Helping Hand Institute of Rehabilitation Sciences, Mansehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai C, Ming G, Ng LY. Development of a clinical prediction rule to identify patients with neck pain who are likely to benefit from home-based mechanical cervical traction. Eur Spine J. 2011 Jun;20(6):912-22. doi: 10.1007/s00586-010-1673-6. Epub 2011 Jan 15. PMID 21240529
- [Background] Sleijser-Koehorst MLS, Coppieters MW, Heymans MW, Rooker S, Verhagen AP, Scholten-Peeters GGM. Clinical course and prognostic models for the conservative management of cervical radiculopathy: a prospective cohort study. Eur Spine J. 2018 Nov;27(11):2710-2719. doi: 10.1007/s00586-018-5777-8. Epub 2018 Oct 16. PMID 30327908